CLINICAL TRIAL: NCT06830785
Title: Effects of Rhythmic Auditory Stimulation on Upper-limb Movements, Function, and Quality of Life in Stroke Patients: A Randomized Controlled Trial
Brief Title: Effects of RAS in Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shu-Mei Wang (Other)
Responsible Party: Sponsor-Investigator, Shu-Mei Wang, Dr., National Taipei University of Nursing and Health Sciences
Organization: National Taipei University of Nursing and Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RAS in stroke patients
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experiment group (Experimental): provision of rhythmic auditory stimulation
  Interventions: Behavioral: rhythmic auditory stimulation incorporated in upper-limb movement training
- Control Group (Active Comparator): no provision of rhythmic auditory stimulation
  Interventions: Behavioral: Upper-limb movement training

INTERVENTIONS:
Behavioral: rhythmic auditory stimulation incorporated in upper-limb movement training — Rhythmic auditory stimulation will be metronome beat sound with different tempi and will be incorporated in upper-limb movement training, which will last for 40 minutes per session, three sessions per week, and a total of 24 sessions.
  Arms: Experiment group
Behavioral: Upper-limb movement training — Upper-limb movement training will last for 40 minutes per session, three sessions per week, and a total of 24 sessions.
  Arms: Control Group

SUMMARY:
The goal of this study is to to examine whether rhythmic auditory stimulation improved movement speed, movement function of executing activities of daily living, and movement recovery of the affected upper limb, as well as quality of life in stroke patients. The main questions it aims to answer are:

* Does rhythmic auditory stimulation improve movement speed in stroke patients?
* Does rhythmic auditory stimulation improve movement function of executing activities of daily living in stroke patients?
* Does rhythmic auditory stimulation improve movement recovery of the affected upper limb in stroke patients?
* Does rhythmic auditory stimulation improve quality of life in stroke patients?

Researchers will compare movement training with the aid of rhythmic auditory stimulation to movement training without the aid of rhythmic auditory stimulation to see if rhythmic auditory stimulation works to improve movement speed, movement function of executing activities of daily living, and movement recovery of the affected upper limb, as well as quality of life in stroke patients.

Participants will:

* Undergo movement tests and fill out questionnaires before and after the movement training program
* Receive movement training for 40 minutes per session and three sessions per week for a total of 24 sessions

ELIGIBILITY:
Inclusion Criteria:

* (1) Diagnosed with either ischaemic or hemorrhagic stroke, and a first-time occurrence;
* (2) A unilateral stroke;
* (3) The onset occurred six months or more prior to the experiment, indicating a chronic stage of stroke;
* (4) The affected upper limb's proximal and distal joints are between Brunnstrom stages four to six, ensuring that the affected limb can execute the upper-limb functional movement training of this study;
* (5) The affected upper limb's Modified Ashworth Scale score is ≤ 2, indicating no significant muscle stiffness (spasticity) in the affected limb;
* (6) A Montreal Cognitive Assessment score of ≥ 24, ensuring comprehension of the instructions given during this study;
* and (7) when we clap hands next to the affected ear of the participant who closes eyes, the participant is able to indicate the sound's source either verbally or through gestures, indicating no complete hearing loss in the affected ear and the ability to receive rhythmic auditory stimulation.

Exclusion Criteria:

* (1) Neurological diseases or medical conditions that affect upper-limb movements or hearing;
* (2) Being participating in other experimental studies related to drug treatment or upper-limb movement therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Nine-Hole Peg Test | Up to 1 week right before the 1st session of the intervention
  A larger value (the recorded time for completing the task) means a slower movement.
Nine-Hole Peg Test | Up to 1 week right after the last session of the intervention
  A larger value (the recorded time for completing the task) means a slower movement.
Box and Block Test | Up to 1 week right before the 1st session of the intervention
  A larger value (the number of blocks) means a faster movement.
Box and Block Test | Up to 1 week right after the last session of the intervention
  A larger value (the number of blocks) means a faster movement.

SECONDARY OUTCOMES:
Jebsen-Taylor Hand Function Test | Up to 1 week right before the 1st session of the intervention
  A larger value (the time for completing the task) of each task means a slower movement.
Jebsen-Taylor Hand Function Test | Up to 1 week right after the last session of the intervention
  A larger value (the time for completing the task) of each task means a slower movement.
the Fugl-Meyer Assessment | Up to 1 week right before the 1st session of the intervention
  A higher value means better movement recovery.
the Fugl-Meyer Assessment | Up to 1 week right after the last session of the intervention
  A higher value means better movement recovery.
the Stroke Impact Scale | Up to 1 week right before the 1st session of the intervention
  A larger value means better quality of life.
the Stroke Impact Scale | Up to 1 week right after the last session of the intervention
  A larger value means better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taipei University of Nursing and Health Sciences, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No